CLINICAL TRIAL: NCT04823143
Title: Natural History of Disease Progression in Individuals With a Confirmed Diagnosis of Disease Caused by Mutation of the Valosin Containing Protein (VCP) Gene
Brief Title: Natural History Study of Patients With VCP-related Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Lindsay Alfano, Principal Investigator, Nationwide Children's Hospital
Other Study IDs: VCP-00-001
Record Dates: First submitted 2021-03-26; First posted 2021-03-30 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: IBMPFD
MeSH Terms: conditions — Inclusion Body Myopathy With Early-Onset Paget Disease And Frontotemporal Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Patients opting in to biosample collection will provide blood, serum, and urine samples for biobanking.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A natural history study to understand the expected progression of disease in patients with confirmed mutations in the VCP gene over 1 year.

DETAILED DESCRIPTION:
This is a single site, prospective natural history study to evaluate the utility of strength, functional, and patient reported outcomes in quantifying disease progression over 1 year in patients with mutations in the VCP gene.

Patients will complete a remote and onsite visits at baseline, a remote visit at 6 months, and then a final remote and onsite visit at 12 months. All strength, functional, and patient reported measures will be completed at each visit to assess reliability, consistency of results across testing environments, and sensitivity to change over time.

Additionally, patients may opt in to provide blood, serum, and urine samples for biobanking.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed mutation in the VCP gene
* Age ≥18 years
* Willing and able to provide informed consent and follow all study procedures

Exclusion Criteria:

* Participation in an interventional clinical trial
* Any concomitant illness or comorbid condition that would interfere with a patient's ability to complete study procedures safely at the discretion of the site PI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients meeting eligibility criteria and able to travel to Columbus Ohio for onsite visits.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2021-03-18 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
100 meter timed test | 12 months
  Patients will complete 100-meter walk/run on a 25-meter course as quickly as possible, safely. The time to complete is recorded.
North Star assessment for limb girdle type dystrophies (NSAD) | 12 months
  A 29-item assessment of functional tasks such as standing, walking, rising from floor, standing on 1 leg, etc. This assessment also includes 2 timed items: rise from floor and 10 meter walk/run. Each task is scored on a 0=unable, 1=completed with compensation, 2=completed without compensation. A total score for all items is recorded.
Timed Up and Go | 12 months
  A patient stands from a chair, walks 3 meters, and returns to sitting in the chair as quickly as possible. The time to complete is recorded.
4 stair climb | 12 months
  Records the fastest time a patient can ascend 4 steps using handrails as needed.
Performance of Upper Limb (PUL) 2.0 | 12 months
  A 22-item assessment of upper extremity tasks such as lifting arms overhead, bringing a cup to mouth, tearing paper, stacking cans, etc. Each task is scored on a 0=unable, 1=completed with compensation, 2=completed without compensation. A total score for all items is recorded.
9 hole peg test | 12 months
  Records the time it takes a patient to place 9 pegs in holes and remove as quickly as possible
Forced Vital Capacity | 12 months
  Records the maximum volume a patient can expire forcefully from their lungs in the seated position.
PROMIS Global Health scale | 12 months
  10 item patient reported measure with questions about a patient's rating of overall health, quality of life, and ability to complete and participate in regular activities.
Neuro-QOL Upper Extremity Function | 12 months
  A patient reported outcome with questions about a person's ability to complete activities of daily living including bathing, dressing, turning a key in a lock, etc
Neuro-QOL Lower Extremity Function (Mobility) | 12 months
  A patient reported outcome with questions about a person's ability to complete mobility activities such as stepping up on curbs, transfers, pushing open doors, etc
Rasch Overall ALS Disability Scale (ROADS) | 12 months
  A 28-item patient reported measure with questions about swallowing, speaking, mobility, and upper extremity tasks.
Neuro-QOL Cognition Function | 12 months.
  A patient reported outcome with questions about a person's regular cognitive ability including reading, thinking, paying attention, and concentrating.
EAT-10 | 12 months
  A 10-item patient-reported assessment with questions related to swallowing function.
Communicative Participation Item Bank (CPIB) | 12 months
  A self-reported measure with questions related to ability to communicate, be understood, and relative difficulty or ease in communicating.
Speech Handicap Index | 12 months
  This patient-reported measure includes questions related to speech functions and abilities.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Alfano, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States